CLINICAL TRIAL: NCT05941533
Title: Infrared Thermal Imaging in Evaluating the Percutaneous Transluminal Angioplasty for Peripheral Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fangge Deng (Other)
Responsible Party: Sponsor-Investigator, Fangge Deng, : Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: IRTIPTA
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Artery Disease (PAD)
Keywords: peripheral artery disease (PAD), infrared thermal imaging (IRTI), percutaneous transluminal angioplasty (PTA)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determination of IRTI (infrared thermal imaging) can be used to evaluate PAD patients with critical limb ischemia with different degrees of lesion.

IRTI can be used to evaluate the foot blood perfusion after percutaneous transluminal angioplasty (PTA) treatment and determine the success rate of surgery.

IRTI can be used as an effective follow-up tool for patients after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Rutherford grade 3, 4, 5, or 6.
* Patients with indications for lower extremity arterial PTA: severe intermittent claudication, rest pain, ulceration or gangrene.
* Patients who required PTA of only one limb (left versus right).

Exclusion Criteria:

* Patients with body temperature above 37 ° C.
* Patients with indications for open surgery.
* Patients requiring major amputation (above the ankle).
* Patients with acute occlusive or embolic limb ischemia.
* Patients with deep venous thrombosis of the lower extremity.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: PAD patients who came to our hospital for diagnosis and treatment were initially selected, and those who met the indications for PTA surgery were finally included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
To determine the validity and reliability of IRTI in assessing foot blood perfusion and surgical success rate after PTA treatment. | up to 15 months
  The different levels of pseudocodes (white, red, pink, yellow, green, blue, and black) represent the corresponding IRTI, corresponding to the color bar from low to high temperature.
  We will measure the average temperature of the dorsum and sole of the foot before and after PTA treatment in the operated and non-operated limbs. Ankle-brachial index (ABI) of the operated and non-operated limbs before and after PTA treatment will also be measured.
  We will analyze the agreement between ABI and foot temperature in the operated and non-operated limbs, as well as the agreement between the change in ABI and foot temperature.

CONTACTS AND LOCATIONS:
Locations (1):
- Fangge Deng, Guangzhou, Guangdong, China